CLINICAL TRIAL: NCT05326464
Title: Tofacitinib: Suppressing Tumor Invasion in Recurrent GBM Patients
Brief Title: Tofacitinib in Recurrent GBM Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Michael Youssef, ASSISTANT PROFESSOR - Neurology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-1029
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tofacitinib 10 mg (Experimental): Participants will take the 10mg Tofacitinib twice daily until evidence of progression, intolerance of treatment, withdrawal of consent, or death.
  Interventions: Drug: Tofacitinib 10mg

INTERVENTIONS:
Drug: Tofacitinib 10mg — 10 mg given orally twice daily until evidence of progression, intolerance of treatment, withdrawal of consent, or death.

SUMMARY:
The purpose of this study is to examine the effects of Tofacitinib in patients with recurrent Glioblastoma.

DETAILED DESCRIPTION:
Once consented and registered, eligible patients will commence Cycle 1 and be assessed on Cycle 1 Day 1. An entire cycle will be 28 days of continuous Tofacitinib dosing. There will be a gap of 18-24 days between the first and subsequent cycles of treatment. The patient will once again be assessed on Cycle 2 Day 1. An interim follow-up will be done after the second cycle, during which the patient will undergo a brain MRI for tumor measurements along with all other assessments. Subsequent cycles will continue as prior, with subject assessments, brain MRI, and toxicity evaluations every 4 weeks. Treatments will stop upon evidence of disease progression, unacceptable toxicity, or if the physician deems it unsafe for the subject to continue in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed GBM (MGMT unmethylated, IDH wild type) at first, second, third, or fourth recurrence after concurrent chemoradiotherapy. Patients with an initial diagnosis of a lower-grade glioma are eligible if a subsequent biopsy determined the progressive tumor to be GBM.
2. Imaging confirmation of first tumor progression or regrowth as defined by the Response Assessment in Neuro-Oncology (RANO) criteria. A minimum of 12 weeks must have elapsed from the completion of radiotherapy to study entry to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progression of disease, unless there is a new lesion outside the radiation field or unequivocal evidence of viable tumor on histopathological sampling.
3. Karnofsky Performance Status (KPS) ≥ 60%.
4. Patients must be willing and able to provide written informed consent and to comply with the study protocol as judged by the investigator.
5. Age ≥ 18 years.
6. Patients must be able to swallow oral medications.
7. For women who are of child-bearing potential and who are sexually active and who are not surgically sterile (absence of ovaries and/or uterus): to use an adequate method of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly) during the treatment period and for at least 6 months after last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. For male patients who are partners of premenopausal women: agreement to use a barrier method of contraception during the treatment period and for at least 6 months after the last dose of study drug.

   7.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
8. Patients who have undergone recent surgery for recurrent or progressive tumor are eligible provided that:

   8.1 Surgery must have confirmed the recurrence.

   8.2 A minimum of 28 days must have elapsed from the day of surgery to study entry. For core or needle biopsy, a minimum of 7 days must have elapsed prior to study entry.

   8.3 Craniotomy or intracranial biopsy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomization.
9. Patients must have recovered (Common Terminology Criteria for Adverse Events CTCAE version 6] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. Minimum times from prior therapies include:

   9.1 Greater than or equal to 28 days elapsed from the administration of any investigational agent.

   9.2 Greater than or equal to 28 days elapsed from the administration of any prior cytotoxic agents, except ≥ 42 days from nitrosoureas. NOTE: Prior treatment with Novo-TTF therapy is allowed at initial diagnosis but must be discontinued prior to study entry.
10. GBMs of the study patients must have EGFR gene amplification, which will be detected by next generation sequencing of tumor tissue from resected sample.
11. Prior use of bevacizumab is allowed, however patient must be off of this medication for 180 days.
12. Patients must have adequate organ and marrow function as defined by the following criteria:

    * ANC ≥1.5 × 10(9)/L
    * Platelets ≥100 × 10(9)/L
    * Hemoglobin ≥8 g/dL
    * Total bilirubin ≤1.5 × ULN Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.

ALT and AST ≤3 × ULN

Exclusion Criteria:

1. Prior treatment with an EGFR or JAK inhibitor.
2. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
3. Patients unable to undergo brain MRI scans with IV gadolinium contrast.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Tofacitinib
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
6. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
7. Prior history of hypertensive crisis, hypertensive encephalopathy, or inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg while on antihypertensive medication).
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant gastrointestinal resection that would preclude adequate absorption of the trial medications.
9. History of another malignancy in the previous 3 years, with a disease-free interval of < 3 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
10. Concurrent use of Bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of the study cohort as defined by RANO criteria. | Up to 2 years after study treatment
  Median progression-free survival from initiation of Tofacitinib until disease progression as defined by the RANO criteria, unacceptable toxicity, withdrawal of consent, or discontinuation from the trial for any other reason.

SECONDARY OUTCOMES:
Overall survival (OS) of the study cohort. | Up to 2 years after study treatment
  Median OS of the study patients from time of study entry until death or lost to follow-up.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | Up to 2 years after study treatment
  Assess safety and tolerability associated with Tofacitinib 5 mg orally twice daily when administered to GBM patients. NCI Common terminology criteria for adverse events (CTCAE v.5) will be used to assess the adverse events.
Tumor response by RANO criteria. | Up to 2 years after study treatment
  Tumor response will be assessed using contrast and non-contrast brain magnetic resonance imaging (MRI) with assessments based on the international criteria proposed by the Response Assessment in Neuro-Oncology (RANO) Working Group, until progression of disease. For patients who do not progress or die, PFS will be censored at the last adequate radiologic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Youssef, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No